CLINICAL TRIAL: NCT02345512
Title: Investigation of Lycra Splinting Garments for Falls and Intellectual Disabilities
Brief Title: Investigating the Clinical and Cost Effectiveness of Lycra Splinting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GlasgowCULycraTrial01
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2018-02

CONDITIONS: Learning Disability
Keywords: Falls
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Falls (Other): Wearing of Lycra splinting garment
  Interventions: Device: Lycra Splinting Garment

INTERVENTIONS:
Device: Lycra Splinting Garment — Wearing of lycra splinting garment for 6 weeks
  Other Names: Dynamic Elastomeric Functional Orthosis

SUMMARY:
People with learning disabilities (LDs) experience high levels of health problems, including cerebral palsy, other problems associated with posture, movement and function, and injury (falls are the commonest cause of injury in this population, and poor balance/coordination are a contributory factor). The aim of this project is to investigate the clinical and cost effectiveness of lycra splinting garments (LSGs), worn to improve posture, movement and function, for adults (16 years and over) with LDs who fall. This project aims to investigate the clinical and cost effectiveness of LSGs to prevent future falls of adults with LDs, to inform practice and guidelines within local and national (National Health Service - NHS) adult services.

Falls and fall injury are a serious problem for people with LDs (people with LDs experience similar rates of falls as the elderly in the general population but at a younger age), whereby interventions are warranted. Lab based 3D movement analysis will be conducted with adults with LDs who fall during two visits to perform simple tasks (e.g. walking) (once prior to being provided with LSG, and once 6 weeks after wearing the LSGs at home).

DETAILED DESCRIPTION:
Adults with Learning Disability who have capacity will be recruited to participate in the Lycra splinting trial via their local physiotherapist. The eligibility criteria is an adult with Learning Disability who has had a fall and who has problems with their balance and/or gait as identified by their local physiotherapist.

The participants will be recruited via participant information sheets. The participants will attend the Glasgow Caledonian University (GCU) gait laboratory to undertake three-dimensional movement analysis; Gaitrite test (the Gaitrite is a commercially available instrumented walkway); and Centre of Pressure testing.

This will take place before prescription of a Lycra splinting garment and a minimum of 6 weeks wear after receiving a Lycra splinting garment.

Analysis of data captured before and after wearing the Lycra splinting garment will take place.

The use-ability of the Lycra splinting garment will also be determined by completion of a user and carer questionnaire and by completion of a questionnaire by their local physiotherapist.

The cost effectiveness of Lycra splinting garments will be analysed by a health statistician within GCU.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a learning disability, and has had a fall within the last 12 months due to a balance or gait issue.

Exclusion Criteria:

* Any participant who does not have capacity to consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Finlayson, PHD, Study Chair — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finlayson J, Crockett J, Shanmugam S, Stansfield B. Lycra splinting garments for adults with intellectual disabilities who fall due to gait or balance issues: a feasibility study. J Intellect Disabil Res. 2018 May;62(5):391-406. doi: 10.1111/jir.12477. Epub 2018 Feb 14. PMID 29441642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via the National Health service physiotherapists in 2 Health Boards.
Groups:
- Lycra Splint: Wearing of Lycra splinting garment
  Lycra Splinting Garment: Wearing of lycra splinting garment for 6 weeks
Period: Overall Study
Arm/Group | Lycra Splint
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Adults with Intellectual Disabilities
Arm/Group | Lycra Splint
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Falls
Description: Self-report fall calendar completed daily during the 6-week intervention period
Time Frame: 6 weeks
Population: Adults with Intellectual Disabilities with gait issues who experienced a fall within the last 12 months
Measure: Mean (Full Range); unit: Falls
Groups:
- All Participants: All participants (no subgroups or arm)
Arm/Group | All Participants
Number analyzed (Participants) | 9
Falls | 3 [0 to 12]

2. Primary Outcome: Center of Pressure Standard Deviation
Description: The standard deviation of the Center of Pressure during quiet standing. The standard deviation of this measure is used as the outcome as it is the dispersion of the location of the centre of pressure that is of interest.
Time Frame: 6 week intervention period
Population: Adults with intellectual disabilities with gait or balance issues who have experienced a fall in previous 12 months
Measure: Mean (Full Range); unit: mm
Groups:
- Baseline: All participants at baseline
- Post Intervention: All participants post intervention
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
mm | 10.6 [5.3 to 24.0] | 9.8 [4.6 to 20.7]

3. Primary Outcome: Walking Speed
Description: The walking speed along a standardised walking mat.
Time Frame: 6 week intervention period
Population: Adults with intellectual disabilities with balance or gait issues who fall
Measure: Mean (Full Range); unit: m/s
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
m/s | 0.593 [0.325 to 0.836] | 0.594 [0.318 to 0.842]

4. Primary Outcome: Step Length
Description: Distance from initial foot contact on one side to initial foot contact on contralateral side.
Time Frame: 6 week intervention period
Population: Adults with intellectual disabilities with gait or balance issues who have fallen in previous 12 months
Measure: Mean (Full Range); unit: m
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
m | 0.402 [0.243 to 0.588] | 0.398 [0.230 to 0.533]

5. Primary Outcome: Base of Support
Description: Width between heel strikes perpendicular to direction of travel
Time Frame: 6 week intervention period
Population: Adults with Intellectual Disabilities with Gait or Balance Issues who Fall
Measure: Mean (Full Range); unit: m
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
m | 0.187 [0.034 to 0.310] | 0.196 [0.066 to 0.322]

6. Primary Outcome: Step Symmetry
Description: The symmetry was calculated as the ratio between the longest and shortest of the left and right step lengths. This provides an indication of the level of symmetry between sides. A score of 1 indicates complete symmetry with values less than one becoming progressively less symmetrical.
Time Frame: 6 week intervention period
Population: Adults with intellectual disabilities with gait or balance issues who have fallen at least once in the previous 12 months
Measure: Mean (Full Range); unit: ratio
Groups:
- Basline: All participants at baseline
Arm/Group | Basline | Post Intervention
Number analyzed (Participants) | 9 | 9
ratio | 0.86 [0.59 to 1.00] | 0.86 [0.62 to 0.98]

7. Primary Outcome: Double Support Time as a Percentage of the Gait Cycle
Description: Percentage of the gait cycle where both feet are on the ground together.
Time Frame: 6 week intervention period
Population: as for outcome 6
Measure: Mean (Full Range); unit: percentage of the gait cycle
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
percentage of the gait cycle | 56.30 [44.21 to 68.74] | 55.80 [42.61 to 66.65]

8. Primary Outcome: Timed Up and Go Test Time
Description: The time taken to complete the Timed Up and Go Test.
Time Frame: 6 week intervention period
Population: as for outcome 6
Measure: Mean (Full Range); unit: s
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 9 | 9
s | 20.68 [9.67 to 40.53] | 19.71 [10.48 to 42.07]

9. Secondary Outcome: Number of Participants That Were Compliant With Lycra Splinting Garment Wear
Description: Survey questions to determine usability (compliance) of lycra splinting garment wear for individuals with intellectual disabilities
Time Frame: 6 week intervention period
Population: adults with intellectual disabilities who had experienced a fall in the last 12 months
Measure: Number; unit: participants
Groups:
- All Participants: All participants together as no subgroups or arms
Arm/Group | All Participants
Number analyzed (Participants) | 9
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the study data collection period which was 6 months.
Arm/Group | Lycra Splint
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lycra Splint (N=11)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) — bruising to buttock area following assistance of putting on Lycra splinting garment.

LIMITATIONS AND CAVEATS:
Small participant numbers did not allow for inferential statistics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No